CLINICAL TRIAL: NCT02351544
Title: Prospective, Multi-Center Evaluation of the Efficacy of Peripheral Trigger Decompression Surgery for Migraine Headaches
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: University of Wisconsin, Madison (Other); Massachusetts General Hospital (Other); University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, Jeffrey Janis, Professor, Ohio State University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015H0024
Record Dates: First submitted 2015-01-21; First posted 2015-01-30 (Estimated); Results first posted 2024-04-22 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Migraine Headaches
MeSH Terms: conditions — Migraine Disorders | interventions — Botulinum Toxins, Type A; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Botulinum toxin (Experimental): Patients in this arm will receive botulinum toxin for migraine headaches
  Interventions: Drug: Botulinum Toxin Type A; Other: Daily headache diary; Other: Migraine Disability Assessment Test (MIDAS); Other: Migraine Work and Productivity Loss Questionnaire (MWPLQ); Other: Migraine-Specific Quality of Life Questionnaire (MSQ)
- Surgery (Experimental): Patients in this arm will receive surgery for migraine headaches
  Interventions: Procedure: Surgery; Other: Daily headache diary; Other: Migraine Disability Assessment Test (MIDAS); Other: Migraine Work and Productivity Loss Questionnaire (MWPLQ); Other: Migraine-Specific Quality of Life Questionnaire (MSQ)

INTERVENTIONS:
Drug: Botulinum Toxin Type A
  Arms: Botulinum toxin
Procedure: Surgery
  Arms: Surgery
Other: Daily headache diary
Other: Migraine Disability Assessment Test (MIDAS)
Other: Migraine Work and Productivity Loss Questionnaire (MWPLQ)
Other: Migraine-Specific Quality of Life Questionnaire (MSQ)

SUMMARY:
According to the peripheral trigger theory of migraine headaches, nociceptive inputs from irritated or compressed cranial nerve branches can lead to neurovascular changes in the brain that cause migraine headaches. Advanced treatments aimed at deactivating the peripheral trigger points can be administered to patients who have failed medical management of migraines. Those accepted advanced treatments include botulinum toxin A injection in order to temporarily paralyze muscles causing nerve compression, and surgery to release those compression points permanently. An advantage of surgery is the ability to release non-muscular causes of nerve compression, such as fascial bands or intersecting arteries.

Botulinum toxin A injection into trigger sites has been shown in multiple studies to be effective at reducing the frequency and severity of migraine headaches, and is a very commonly administered treatment for refractory migraines. It is approved by the FDA for the treatment of chronic migraines.

Similarly, surgical decompression of trigger sites has previously been shown to have superior clinical outcomes to medical management, through a randomized, blinded controlled-trial performed at Case Western Reserve in 2009. Patients either received actual decompression of the trigger sites, or sham surgery (exposure and visualization of the trigger sites, without decompression). At one-year follow-up, the group who underwent actual surgery demonstrated a statistically higher proportion with significant improvement in their migraines (83.7% vs. 57.7%, p=0.014), and with complete elimination of their migraines (57.1% vs. 3.8%, p<0.001). Several other reports have confirmed the good clinical outcomes of surgery demonstrated in this trial, and surgical decompression is now commonly performed by several surgeons around the United States.

Prognostic factors predicting the success of surgical decompression in migraine headache treatment include older age of migraine onset, visual symptoms/aura, and 4-site decompression. Factors predicting failure of surgery include excessive operative blood loss, and surgery on only one or two trigger sites.

One criticism of the studies on peripheral trigger decompression surgery for migraines has been that most of the results have originated from the same institution (Case Western Reserve), and from the same author (Guyuron). While several studies at other institutions have demonstrated positive outcomes of peripheral trigger decompression, these have only included a small number of patients.

In addition, the sham surgery randomized-controlled trial has been criticized for not clarifying any prior treatments that patients had undergone before peripheral trigger deactivation, and for not showing how medication use patterns changed after surgery. Another criticism of that study was the fact that patients were examined by neurologists before the study but not after the study, and that surgery was performed on some patients with episodic migraines, who are known to not benefit from botulinum toxin. It is unclear what migraine types are most likely to benefit from surgical decompression.

The investigators' goal is to perform a multi-center, prospective trial to demonstrate the effectiveness of peripheral trigger decompression in the treatment of migraine headaches, which would address the criticisms mentioned above. The main aim is to demonstrate that the positive results demonstrated by Guyuron et al are reproducible at other institutions and by other surgeons using similar techniques on different patient populations.

ELIGIBILITY:
Inclusion Criteria:

* Patients with migraines related to a trigger site at the location of a branch of a cranial nerve (frontal, temporal, occipital)
* Patients with chronic migraine (≥15 days per month) as dictated by the FDA indication for botulinum, and as diagnosed by a board-certified neurologist
* Patients with episodic migraines

  * Those patients are included because there is no consensus whether surgical decompression is effective for chronic migraines only, or for chronic and episodic migraines. One of the goals of this trial is to determine this.
* Patients who respond to diagnostic botulinum toxin injection or to a diagnostic anesthetic block
* Patients who have failed 2 of 3 classes of preventative migraine medications

Exclusion Criteria:

* Patients deemed by the authors or the neurologist to not have migraine headaches, but an alternative diagnosis
* Patients with systemic conditions that make them poor candidates for surgery (coronary artery disease, uncontrolled diabetes mellitus, etc…)
* Patients with migraines related to inferior turbinate hypertrophy or septal deviation
* Patients with a frontal, temporal or occipital trigger point who do not respond to a diagnostic botulinum toxin injection or to a diagnostic anesthetic block
* Hypersensitivity to any botulinum toxin preparation or to any of the components in the formulation
* Infection at the proposed injection site for botulinum
* Patients with trigger points at minor trigger sites (lesser occipital nerve, third occipital nerve)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2022-06 (Actual); Study Completion 2022-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Peled Plastic Surgery, San Francisco, California
  - Premier Plastic Surgery of Kansas City, Olathe, Kansas
  - Massachusetts General Hospital, Boston, Massachusetts
  - Neuropax Clinic, St Louis, Missouri
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - The University of Wisconsin-Madison, Madison, Wisconsin

RESULTS

PARTICIPANT FLOW:
Groups:
- Botulinum Toxin: Patients in this arm will receive botulinum toxin for migraine headaches
  Botulinum Toxin Type A
  Daily headache diary
  Migraine Disability Assessment Test (MIDAS)
  Migraine Work and Productivity Loss Questionnaire (MWPLQ)
  Migraine-Specific Quality of Life Questionnaire (MSQ)
- Surgery: Patients in this arm will receive surgery for migraine headaches
  Surgery
  Daily headache diary
  Migraine Disability Assessment Test (MIDAS)
  Migraine Work and Productivity Loss Questionnaire (MWPLQ)
  Migraine-Specific Quality of Life Questionnaire (MSQ)
Period: Overall Study
Arm/Group | Botulinum Toxin | Surgery
Started | 11 | 33
Completed | 11 | 33
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Botulinum Toxin | Surgery | Total
Number analyzed (Participants) | 11 | 33 | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 33 | 44
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.1 (14.3) | 43.8 (12.7) | 43 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 29 | 39
  Male | 1 | 4 | 5
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 11 | 33 | 44

OUTCOME MEASURES:

1. Primary Outcome: Migraine Headache Index (MHI) at 1 Year
Description: MHI is a numerical value calculated by multiplying the severity (1-10 numerical rating scale), duration (fraction of 24 h), and frequency (days per month) of migraine headaches. The lower the value the lower migraine severity reported is. The index range is minimum 0.00 to maximum 300.00.
Time Frame: 1 year postoperatively
Population: Patients enrolled and analyzed in each group for this outcome measure.
Measure: Mean (95% Confidence Interval); unit: index score
Arm/Group | Botulinum Toxin | Surgery
Number analyzed (Participants) | 11 | 12
index score | 7.81 [2.44 to 21.53] | 3.73 [0.94 to 10.53]

2. Primary Outcome: Migraine Headache Index (MHI) at 2 Years
Description: as for outcome 1
Time Frame: 2 years postoperatively
Population: patients enrolled and analyzed in each group for this outcome measure.
Measure: Mean (95% Confidence Interval); unit: index score
Arm/Group | Botulinum Toxin | Surgery
Number analyzed (Participants) | 10 | 10
index score | 61.12 [34.23 to 108.53] | 5.54 [1.52 to 15.94]

3. Primary Outcome: Migraine Headache Index (MHI) at 2.5 Years
Description: as for outcome 1
Time Frame: 2.5 years postoperatively
Population: participants and enrolled and analyzed for this outcome measure
Measure: Mean (95% Confidence Interval); unit: index score
Arm/Group | Botulinum Toxin | Surgery
Number analyzed (Participants) | 3 | 2
index score | 8.74 [2.69 to 24.72] | 1.28 [0.00 to 13.70]

4. Secondary Outcome: Migraine Disability Assessment Test (MIDAS) Score at 1 Year
Description: MIDAS questionnaire was developed to quantify the effect of headaches on patients' daily functionality in the past 3 months. It consists of five questions related to paid work or school, household work, and leisure time. A total score of 0-5 corresponds to little or no disability, 6-10 points refers to mild disability, 11-20 points mean moderate disability, and more than 21 points represent severe disability (MIDAS total). For MIDAS total, the higher the numeric response, the greater the overall impact of MH. The minimum score is 0.00 and the maximum score is 90.00.
Time Frame: 1 year postoperatively
Population: participants enrolled and analyzed in this outcome measure at this time point
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Botulinum Toxin | Surgery
Number analyzed (Participants) | 11 | 28
units on a scale | 17.05 [6.27 to 43.82] | 8.84 [4.62 to 16.22]

5. Secondary Outcome: Migraine Disability Assessment Test (MIDAS) Score at 2 Years
Description: as for outcome 4
Time Frame: 2 years postoperatively
Population: participants enrolled and analyzed for this outcome at this timepoint
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Botulinum Toxin | Surgery
Number analyzed (Participants) | 10 | 24
units on a scale | 10.84 [3.62 to 29.33] | 7.60 [3.76 to 14.54]

6. Secondary Outcome: Migraine Disability Assessment Test (MIDAS) Score at 2.5 Years
Description: as for outcome 4
Time Frame: 2.5 years postoperatively
Population: participants enrolled and analyzed in the outcome measure at the timepoint
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Botulinum Toxin | Surgery
Number analyzed (Participants) | 3 | 10
units on a scale | 10.25 [1.48 to 50.08] | 10.55 [3.98 to 25.79]

7. Secondary Outcome: Migraine Work and Productivity Loss Questionnaire (MMWPLQ) Score at 1 Year
Description: MWPLQ has nine questions that evaluate the impact of migraine and migraine therapy on paid work and productivity loss. Question #7 from the MWPLQ (MWPLQ7) was the most frequently and consistently answered with meaningful responses and did not depend on questions #1-6, 8-9. Therefore, MWPLQ7 was analyzed independently, and the remaining questions were not included in the final analysis. Question #7 assesses the difficulty of 18 work-related activities caused by the most recent MH or migraine headache treatment. Each item in question 7 has the following options: 0 ('no difficulty'), 1 ('a slight amount'), 2 ('some'), 3 ('quite a bit'), 4 ('a great deal'), 5 ('so much difficulty, could not do at all'), and 6 ('does not apply to my work'). To quantify difficulty, a total sum score of these 18 items including only options 0 to 5 is obtained. A higher MWPLQ7 summed score reveals a higher (worse) effect of MH on work and productivity. The minimum is 0.00 and the maximum is 90.00
Time Frame: 1 year postoperatively
Population: participants enrolled and analyzed for this outcome measure at this timepoint
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Botulinum Toxin | Surgery
Number analyzed (Participants) | 10 | 16
units on a scale | 40.44 [20.73 to 78.03] | 16.03 [9.34 to 27.06]

8. Secondary Outcome: Migraine Work and Productivity Loss Questionnaire (MMWPLQ) Score at 2 Years
Description: as for outcome 7
Time Frame: 2 years postoperatively
Population: participants enrolled and analyzed for this outcome measure at this timepoint
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Botulinum Toxin | Surgery
Number analyzed (Participants) | 9 | 11
units on a scale | 34.68 [17.21 to 68.87] | 7.63 [3.82 to 14.41]

9. Secondary Outcome: Migraine Work and Productivity Loss Questionnaire (MMWPLQ) Score at 2.5 Years
Description: as for outcome 7
Time Frame: 2.5 years postoperatively
Population: participants enrolled and analyzed for this outcome measure during this timepoint
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Botulinum Toxin | Surgery
Number analyzed (Participants) | 3 | 7
units on a scale | 26.62 [8.55 to 78.91] | 9.79 [4.30 to 20.99]

10. Secondary Outcome: Migraine-Specific Quality of Life Questionnaire (MSQ) Score at 1 Year
Description: MSQ is a 14-item questionnaire that evaluates the long-term perceived impact of MH on health-related quality of life over the past 4 weeks. Responses per item include a 6-point scale: 'none of the time,' 'a little bit of the time,' 'some of the time,' 'a good bit of the time,' 'most of the time,' and 'all of the time.' Each option is assigned a score of 1 to 6, respectively. Each domain is scored independently as a sum of items and rescaled from a 0 to 100 scale, with higher scores indicating better quality of life. MSQ survey was analyzed in totality. A higher MSQ sum reflects patient improvement in quality of life. The minimum is 0.00 and the maximum is 270.00.
Time Frame: 1 year postoperatively
Population: participants enrolled and analyzed during this timepoint for this outcome
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Botulinum Toxin | Surgery
Number analyzed (Participants) | 11 | 30
units on a scale | 55.05 [31.62 to 95.30] | 60.61 [43.41 to 84.47]

11. Secondary Outcome: Migraine-Specific Quality of Life Questionnaire (MSQ) Score at 2 Years
Description: as for outcome 10
Time Frame: 2 years postoperatively
Population: participants enrolled and analyzed for this outcome measure at this timepoint
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Botulinum Toxin | Surgery
Number analyzed (Participants) | 10 | 26
units on a scale | 61.12 [34.23 to 108.53] | 43.42 [30.27 to 62.10]

12. Secondary Outcome: Migraine-Specific Quality of Life Questionnaire (MSQ) Score at 2.5 Years
Description: as for outcome 10
Time Frame: 2.5 years postoperatively
Population: participants enrolled and analyzed at this outcome measure at this timepoint
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Botulinum Toxin | Surgery
Number analyzed (Participants) | 3 | 13
units on a scale | 74.30 [26.08 to 208.37] | 37.73 [22.66 to 62.40]

ADVERSE EVENTS:
Time Frame: 2.5 years
Arm/Group | Botulinum Toxin | Surgery
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/33
Other Adverse Events (participants affected / at risk) | 0/11 | 0/33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2014-02-16): https://cdn.clinicaltrials.gov/large-docs/44/NCT02351544/Prot_000.pdf
  • Statistical Analysis Plan (2014-02-16): https://cdn.clinicaltrials.gov/large-docs/44/NCT02351544/SAP_001.pdf